CLINICAL TRIAL: NCT07010588
Title: Comparison of ultraSound, Abbreviated MRI witH and Without HBP aS mOdalities for HCC suRveillance in patienTs With High Risk: a Multi-centers, Randomized Controlled Open-label Trial
Brief Title: Comparison of ultraSound, Abbreviated MRI witH and Without HBP aS mOdalities for HCC suRveillance in patienTs With High Risk
Acronym: SHORT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: National Research Institute for Family Planning (Unknown)
Responsible Party: Principal Investigator, Wang Yi, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2025-Z-43
Record Dates: First submitted 2025-05-19; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma (HCC); Magnetic Resonance Imaging (MRI); Randomized Controlled Trial
Keywords: Hepatocellular carcinoma; magnetic resonance imaging; surveillance
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): After being enrolled, the participants will undergo a liver US examination and a serum AFP test every six months. For those participants who are suspected HCC, an enhanced abdominal CT or enhanced MRI will be performed for confirmation. If the imaging suggests HCC, the research subject will be removed from the group and enter the clinical routine diagnosis and treatment process. If there is no evidence of HCC, the subject will continue to be followed up as planned. Finally, at the end of the 18-month follow-up period, a routine enhanced abdominal CT/MRI will be carried out to confirm the presence of HCC. After the completion of 18 months surveillance, researchers will continue long-term follow-up for another 24 months.
- Non-contrast abbreviated MRI group (Experimental): After the participants are enrolled, a serum AFP test and a NC-AMRI examination including T2-weighted imaging (T2WI) and diffusion-weighted imaging (DWI) will be conducted at the 6th month. A liver US examination and a serum AFP test will be carried out at the 12th month. A serum AFP test and a NC-AMRI examination will be performed at the 18th month. For those participants who are suspected HCC, an enhanced abdominal CT or enhanced MRI will be performed for confirmation. If the imaging suggests HCC, the research subject will be removed from the group and enter the clinical routine diagnosis and treatment process. If there is no evidence of HCC, the subject will continue to be followed up as planned. Finally, at the end of the 18-month follow-up period, a routine enhanced abdominal CT/MRI will be carried out to confirm the presence of HCC. After the completion of 18 months surveillance, researchers will continue long-term follow-up for another 24 months.
  Interventions: Device: non-contrast abbreviated MRI (NC-AMRI)
- Enhanced abbreviated MRI group (Experimental): After the participants are enrolled, a serum AFP test and a E-AMRI examination (using gadoxetic acid disodium) including T2WI, DWI and hepatobiliary phase (HBP) images will be conducted at the 6th month. A liver US examination and a AFP test will be carried out at the 12th month. A serum AFP test and a E-AMRI examination will be performed at the 18th month. For those participants who are suspected HCC, an enhanced abdominal CT or enhanced MRI will be performed for confirmation. If the imaging suggests HCC, the research subject will be removed from the group and enter the clinical routine diagnosis and treatment process. If there is no evidence of HCC, the subject will continue to be followed up as planned. Finally, at the end of the 18-month follow-up period, a routine enhanced abdominal CT/MRI will be carried out to confirm the presence of HCC. After the completion of 18 months surveillance, researchers will continue
  Interventions: Device: enhanced abbreviated MRI (E-AMRI)

INTERVENTIONS:
Device: non-contrast abbreviated MRI (NC-AMRI) — Non-contrast abbreviated MRI (NC-AMRI) examination include T2-weighted imaging (T2WI) and diffusion-weighted imaging (DWI), which takes 10 minutes approximately.
  Arms: Non-contrast abbreviated MRI group
Device: enhanced abbreviated MRI (E-AMRI) — E-AMRI examination (using gadoxetic acid disodium) including T2-weighted imaging (T2WI) and diffusion-weighted imaging (DWI)and hepatobiliary phase (HBP) images, which takes 15 minutes approximately.
  Arms: Enhanced abbreviated MRI group

SUMMARY:
Active surveillance in high-risk hepatocellular carcinoma (HCC) populations enables early detection of tumors. The currently recommended monitoring protocol involves biannual serum alpha-fetoprotein (AFP) testing combined with liver ultrasound (US) examinations. However, conventional US demonstrates limited sensitivity in detecting early-stage HCC lesions.

MRI demonstrates high sensitivity in monitoring cirrhotic patients, but prolonged scanning time limits its routine clinical application. Several abbreviated MRI protocols have been developed for HCC detection, aiming to reduce acquisition time while improving early-stage HCC diagnostic accuracy.

The main question this clinical trial aims to answer is:

Can non-contrast abbreviated MRI (NC-AMRI) and enhanced abbreviated MRI (E-AMRI) detect more early-stage HCC lesions compared to US-based screening? Researchers will randomly divide the participants into three groups in a 1:1:1 ratio, with different surveillance strategies, focused on early HCC detection rates.

DETAILED DESCRIPTION:
Active surveillance in high-risk hepatocellular carcinoma (HCC) populations enables early detection of tumors. Current guidelines recommend biannual AFP testing with liver ultrasound (US), but US has suboptimal sensitivity for early HCC detection.

MRI, while highly sensitive for monitoring cirrhotic patients, is limited in routine use due to long scan times.. Several abbreviated MRI protocols have been developed for HCC detection, aiming to reduce acquisition time while improving early-stage HCC diagnostic accuracy.

This is a multicenter, randomized controlled, open-label clinical trial targeting individuals at high risk for HCC, with a planned enrollment of 1,389 participants.

This trial aims to evaluate the effectiveness of three surveillance strategies-US, non-contrast abbreviated MRI (NC-AMRI; T2WI/DW sequences ) and enhanced abbreviated MRI (E-AMRI; using gadoxetic acid disodium with T2WI/DWI/HBP sequences)-in the active monitoring of HCC in high-risk populations.

Researchers will randomly assign participants (1:1:1) to three surveillance arms, followed by a 24-month long-term follow-up after the initial 18-month monitoring. The study includes 18 months of active surveillance and 24 months of extended follow-up.

The surveillance protocols of three groups:

1. Control: Biannual US + AFP;
2. NC-AMRI: Alternating NC-AMRI (T2WI/DWI) and US at 6/18 months;
3. E-AMRI: Alternating E-AMRI (T2WI/DWI/HBP with gadoxetic acid) and US at 6/18 months.

All the participants will be followed up every 6 months according to the above-mentioned grouping and follow-up contents. For those participants who are suspected HCC, an enhanced abdominal CT or enhanced MRI will be performed for confirmation. If the imaging suggests HCC, the research subject will be removed from the group and enter the clinical routine diagnosis and treatment process. If there is no evidence of HCC, the subject will continue to be followed up as planned. Finally, at the end of the 18-month follow-up period, a routine enhanced abdominal CT/MRI will be carried out to confirm the presence of HCC.

The primary focus of the clinic trial is the the early-stage (BCLC 0+A stage) HCC detection rate at 18th month post-enrollment, with pairwise comparisons among the three strategies.

χ² tests will compare detection rates, sensitivity, and specificity; Kaplan-Meier analysis with log-rank tests will evaluate survival. Survival analysis will include all HCC cases diagnosed in the study.

ELIGIBILITY:
Inclusion criteria

* According to the Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2024 Edition) from department of medical administration, nation health commission of the People's Republic of China, with any one of the following high-risk factors for liver cancer: hepatitis B and/or C virus infection, excessive alcohol consumption, hepatic steatosis or metabolic dysfunction-associated liver disease, dietary exposure to aflatoxin B1, liver cirrhosis from other causes, or a family history of liver cancer, and an aMAP score (age⁃male⁃albi⁃platelets score) of 60-100 points.
* Liver disease patients with no evidence of suspected liver cancer in any imaging examination (liver US, contrast-enhanced CT, or contrast-enhanced MRI) within the past six months.
* Signed informed consent form.

Exclusion Criteria:

* History of previous liver cancer diagnosis.
* Baseline screening at enrollment diagnosed with liver cancer.
* Child-Pugh score ≥ 10 (class C).
* History of other malignant tumors.
* Pregnant or lactating women.
* Clinically diagnosed severe heart/lung disease or uncontrolled comorbidities, with investigator-judged life expectancy < 2 years.
* Glomerular filtration rate < 50 mL/min.
* Inability to undergo (enhanced) MRI due to contraindications or relative contraindications.
* Poor compliance or unsuitability for the clinical trial as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1389 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
the early-stage and very early-stage HCC detection rate | at 18th month
  The primary outcome measure is the proportion of early-stage (BCLC 0+A stage) HCC diagnoses at 18th month, when a routine enhanced abdominal CT/MRI will be carried out to confirm the presence of HCC.

SECONDARY OUTCOMES:
18th month mortality rate in HCC patients | at 18th month
  Number of deaths/population of HCC patients*100%
18th month survival rate in HCC patients | at 18th month
  Number of survivals/population of HCC patients*100%
18th median survival time in HCC patients | at 18th month
  Survival analysis will be performed using the Kaplan-Meier method for patients who developed HCC during the study period
Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV). | at 18th month
  Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).
the incremental cost-effectiveness ratio (ICER) | at 18th month
  ICER (NC-AMRI)=(Total costs of NC-AMRI group)-(Total Costs of control group) / (Number of early-stage HCC patients detected in NC-AMRI group)- (Number of early-stage HCC patients detected in control group) .
  ICER (E-AMRI)=(Total costs of E-AMRI group)-(Total Costs of control group) / (Number of early-stage HCC patients detected in E-AMRI group)- (Number of early-stage HCC patients detected in control group).
  Total costs should include:
  * Direct medical costs (Screening/diagnostic procedures e.g. MRI, blood tests)
  * Direct non-medical costs (Transportation)
  * Indirect costs
  A below-threshold ICER confirms the cost-effectiveness of the new intervention.
Patient compliance to the study protocol | at 18th month
  (Number of enrolled participants) - (Number of loss to follow-up cases)/(Number of enrolled participants)
Patient acceptability to the study protocol | at 18th month
  Collect data by conducting a questionnaire survey among participants
early and very early-stage HCC detection at 42th month | at 42th month
  Proportion of early and very early-stage HCC detection.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Wang, Professor, Study Chair — Peking University People's Hospital
Locations (12):
- China (12):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Handan Central Hospital, Handan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - China-Japan Union Hospital, Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xishuangbanna Dai Autonomous Prefecture, Xishuangbanna Dai Autonomous Prefecture, Yunnan

REFERENCES:
- [Background] Kim SY, An J, Lim YS, Han S, Lee JY, Byun JH, Won HJ, Lee SJ, Lee HC, Lee YS. MRI With Liver-Specific Contrast for Surveillance of Patients With Cirrhosis at High Risk of Hepatocellular Carcinoma. JAMA Oncol. 2017 Apr 1;3(4):456-463. doi: 10.1001/jamaoncol.2016.3147. PMID 27657493
- [Background] Yu NC, Chaudhari V, Raman SS, Lassman C, Tong MJ, Busuttil RW, Lu DS. CT and MRI improve detection of hepatocellular carcinoma, compared with ultrasound alone, in patients with cirrhosis. Clin Gastroenterol Hepatol. 2011 Feb;9(2):161-7. doi: 10.1016/j.cgh.2010.09.017. Epub 2010 Oct 1. PMID 20920597
- [Background] Tzartzeva K, Obi J, Rich NE, Parikh ND, Marrero JA, Yopp A, Waljee AK, Singal AG. Surveillance Imaging and Alpha Fetoprotein for Early Detection of Hepatocellular Carcinoma in Patients With Cirrhosis: A Meta-analysis. Gastroenterology. 2018 May;154(6):1706-1718.e1. doi: 10.1053/j.gastro.2018.01.064. Epub 2018 Feb 6. PMID 29425931
- [Background] Colli A, Fraquelli M, Casazza G, Massironi S, Colucci A, Conte D, Duca P. Accuracy of ultrasonography, spiral CT, magnetic resonance, and alpha-fetoprotein in diagnosing hepatocellular carcinoma: a systematic review. Am J Gastroenterol. 2006 Mar;101(3):513-23. doi: 10.1111/j.1572-0241.2006.00467.x. PMID 16542288
- [Background] Simmons O, Fetzer DT, Yokoo T, Marrero JA, Yopp A, Kono Y, Parikh ND, Browning T, Singal AG. Predictors of adequate ultrasound quality for hepatocellular carcinoma surveillance in patients with cirrhosis. Aliment Pharmacol Ther. 2017 Jan;45(1):169-177. doi: 10.1111/apt.13841. Epub 2016 Nov 8. PMID 27862091
- [Background] Wong LL, Reyes RJ, Kwee SA, Hernandez BY, Kalathil SC, Tsai NC. Pitfalls in surveillance for hepatocellular carcinoma: How successful is it in the real world? Clin Mol Hepatol. 2017 Sep;23(3):239-248. doi: 10.3350/cmh.2017.0008. Epub 2017 Jul 14. PMID 28706177